CLINICAL TRIAL: NCT05239260
Title: Impact of Fluid Status on Liver Elastography and T1-mapping Results in Patients Undergoing CMR.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Andreas Kammerlander, MD Phd, Medical University of Vienna
Other Study IDs: Liver-T1-CMR-2575
Record Dates: First submitted 2022-02-05; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: NAFLD/MAFLD; Liver Fibrosis; CMR
Keywords: NAFLD; CMR
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CMR — CMR
  Other Names: Fibroscan; Body composition monitor

SUMMARY:
Correlation between CMR T1-times, liver T1-times, fibroscan and fluid status to identify the correlation and pathogenesis of liver disease in patients with heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Referred for Cardiovascular Magnetic Resonance Imaging

Exclusion Criteria:

* Non-compatible Devices

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All-comer cohort referred for Cardiovascular Magnetic Resonance Imaging
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Impact of fluid status on liver elastography and T1-times | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kammerlander, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University Vienna, Vienna, Austria